CLINICAL TRIAL: NCT00848575
Title: A Preliminary Study Utilizing a Flexible Endoscope for Pelvic Culdoscopy
Acronym: Culdo
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 99075
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Diagnostic or Therapeutic Laparoscopy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1 - Device: The principal Investigator and sub-investigators of this study will identify potential participants that attend the gynecologic oncology or gynecology clinics of UAMS. These subjects will have been scheduled for diagnostic or therapeutic laparoscopy. Based on the Inclusion Criteria and Exclusion Criteria of this study, women who are eligible for the study will be approached to participate.
  Interventions: Device: Flexible Endoscope

INTERVENTIONS:
Device: Flexible Endoscope

SUMMARY:
The culdoscopic approach will allow for equal or better visualization of female pelvic structures

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 18 to 70 years old
* Ability to understand and give informed consent
* Scheduled for diagnostic or therapeutic laparoscopy for a clinical indication
* Presence of a uterus and at least one ovary at the initiation of the procedure

Exclusion Criteria:

* Documented culdesac mass
* Inability to tolerate anesthesia
* Documentation of positive urine pregnancy test
* History of prior pelvic radiation
* Scheduled for emergency laparoscopy
* Any other medical or psychiatric condition that, in the opinion of the investigative team, will interfere with the ability of the participant to safely complete the study
* History of significant non-compliance with previous therapy or unwillingness to return for follow up visits
* Prior hysterectomy and/or bilateral salpingo-oophorectomy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from among women attending the gynecologic clinics or gynecologic oncology clinic of UAMS. Subjects from all races and ethnicities may participate. No children (aged <18 years) are to be enrolled.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Visualization of female pelvic structures using a flexible endoscope and a standard laparoscope will be compared. | 02/2010

SECONDARY OUTCOMES:
Complications related to the procedures will be recorded and, if possible, attributed to one of the two techniques. If feasible, a comparison will be made between complications attributable to each approach. | 02/2010

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Burnett, MD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States